CLINICAL TRIAL: NCT05771857
Title: Obesity: an Underappreciate Risk Factor for Severe Form of COVID-19: Retrospective Cohort Study of 415 Cases
Brief Title: Obesity: an Underappreciate Risk Factor for Severe Form of COVID-19
Status: Completed | Type: Observational
Sponsor: Mohammed VI University Hospital (Other)
Responsible Party: Principal Investigator, Younes Oujidi, Doctor, Mohammed VI University Hospital
Other Study IDs: Service anesthesie Reanimation
Record Dates: First submitted 2023-03-14; First posted 2023-03-16 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: COVID-19 Pandemic; Obesity
MeSH Terms: conditions — COVID-19; Obesity | interventions — Adiposity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Obesity — the objective of identifying the epidemiological profil of the patients, as well as, the clinical, radiological and prognosis of obese patients with covid 19

SUMMARY:
Our study has the objective of identifying the epidemiological profil of the patients, as well as, the clinical, radiological and prognosis of obese patients with covid 19.

DETAILED DESCRIPTION:
Introduction: COVID 19 pandemic continues to progress with a considerable mortality and morbidity throughout the world since its emergence in December 2019. Many studies were conducted to identify the predictive factors of mortality of those infected with the virus. The previous studies noticed that obesity seems to be associated with severe form of respiratory distress syndrome. Our study has the objective of identifying the epidemiological profil of the patients, as well as, the clinical, radiological and prognosis of obese patients with covid 19.

Methods: investigators led a retrospective monocentric, descriptive and analytic study, in the department of anesthesia and intensive care unit of the university hospital of Mohamed VI Oujda, in Morocco, from March 2020 to October 2021, including all the patients tested positive for the infection.

ELIGIBILITY:
Inclusion Criteria:

* All patients presenting an infection with SARS-CoV-2 that were hospitalized in the intensive care unit.

Exclusion Criteria:

* None

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: investigators have included all the patients presenting an infection with SARS-CoV-2 (1069 patients) diagnosed following the regarding of the world health organization (WHO), confirmed by a PCR of a nasopharyngeal swap, or highly suspected images on thoracic CT scans, that were hospitalized in the intensive care unit.
Sampling Method: Non-Probability Sample
Enrollment: 415 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Obesity: An underappreciate risk factor for severe form of COVID-19: Retrospective cohort study of 415 cases | in all the 22 mounths
  Is obesity a predictive factor of need of intensive care, in addition to the mortality of covid 19?
Risk factor for severe form of COVID-19 | in all the 22 mounths
  identify the epidemiological profil of the patients, as well as, the clinical, radiological and prognosis of obese patients with covid 19.

CONTACTS AND LOCATIONS:
Locations (1):
- younes Oujidi, Berkane, Morocco

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Simonnet A, Chetboun M, Poissy J, Raverdy V, Noulette J, Duhamel A, Labreuche J, Mathieu D, Pattou F, Jourdain M; LICORN and the Lille COVID-19 and Obesity study group. High Prevalence of Obesity in Severe Acute Respiratory Syndrome Coronavirus-2 (SARS-CoV-2) Requiring Invasive Mechanical Ventilation. Obesity (Silver Spring). 2020 Jul;28(7):1195-1199. doi: 10.1002/oby.22831. Epub 2020 Jun 10. PMID 32271993
- [Background] Gao F, Zheng KI, Wang XB, Sun QF, Pan KH, Wang TY, Chen YP, Targher G, Byrne CD, George J, Zheng MH. Obesity Is a Risk Factor for Greater COVID-19 Severity. Diabetes Care. 2020 Jul;43(7):e72-e74. doi: 10.2337/dc20-0682. Epub 2020 May 14. No abstract available. PMID 32409499
- [Background] Yu W, Rohli KE, Yang S, Jia P. Impact of obesity on COVID-19 patients. J Diabetes Complications. 2021 Mar;35(3):107817. doi: 10.1016/j.jdiacomp.2020.107817. Epub 2020 Nov 26. PMID 33358523